CLINICAL TRIAL: NCT07268469
Title: Interception of Minimal Residual Disease in Solid Malignancies
Brief Title: Minimal Residual Disease in Solid Malignancies
Acronym: IMRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UID 5046; L2-397 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer; Non Small Cell Lung Cancer; Prostate Cancer; High Grade Serous Ovarian Cancer; Gastric Cancer
Keywords: ctDNA
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ctDNA detection (Other)
  Interventions: Biological: ctDNA detection

INTERVENTIONS:
Biological: ctDNA detection — a baseline plasma sample will be collected at the time of surgery and prior to the start of adjuvant treatments forassessing the detection of ctDNA.

SUMMARY:
The IMRD study is a single-centre, prospective observational study which will investigate the rate of ctDNA (circulating tumor DNA) detection from the start of adjuvant therapy following curative-intent surgery. The study will include patients of age 18 years old or older, who provided informed consent. Eligible patients are affected by one of the following non-metastatic resected tumors: i) breast cancer (BC), ii) non-oncogene addicted (EGFR/ALK-wild type) non-small-cell lung cancer (NSCLC), iii) high-risk and very high-risk prostate cancer, iv) high-grade serous ovarian cancer (HGSOC), and v) gastric cancer. Eligible patients will undergo surgery and receive adjuvant treatment(s) as per standard guidelines. Patients who underwent neoadjuvant treatments and had a complete pathological response (i.e., no residual tumor at surgery following neoadjuvant treatments) will not be eligible for the present study.

During adjuvant treatment and following its conclusion, patients will be subjected to instrumental monitoring, as per standard guidelines and clinical practice. For eligible patients, a baseline plasma sample will be collected at the time of surgery (feasibility window) and prior to the start of adjuvant treatments (not prior to 28 from the date of surgery) for assessing the detection of ctDNA. Afterwards, plasma samples will be collected at 3, 6 and 9 months from the start of postoperative adjuvant treatments. For patient specific monitoring, a tumor-informed targeted sequencing panel, using tumor-specific mutations detected with WES, will be employed to gather the most sensitive diagnostic platforms, mitigating the risk of negative cases. At 6 months or upon positive ctDNA detection, either a thoracic-abdominal-pelvic or total-body CT scan will be performed to exclude the presence of overt metastatic disease. All patients included in the study will be monitored with longitudinal ctDNA assessment until one-year or follow-up or until the radiological detection of metastatic disease, whichever will occur first. Additional follow-up will be carried outside the IMRD study and will follow standard clinical protocols and schedules. Being an observational study, no treatment intervention will be applied as per protocol based on the detection or absence of ctDNA. For conducting exploratory analyses, the primary tumors will be retrieved and subjected to WES, and the study will aim to detect molecular tumor variables associated with a lack of ctDNA clearance following curative-intent treatment interventions.

The study will be conducted in 2 phases. The first phase aims at verifying the feasibility and sustainability of such approach, based on the identification of at least 15% positive patients. This phase is predicted to be completed within 2 years, and is the object of the present application. If the first endpoint is achieved, we will expand the study to include the co-primary endpoint, which aims at estimating the fraction of patients with persistent ctDNA 6 months post-surgery despite adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Age ≥18 years
* Eligibility for potentially-curative surgery, regardless of previous neoadjuvant/pre-operative systemic treatment
* Completed adequate pre-surgical staging procedures as per standard clinical practice
* Diagnosis of one of the following:
* Clinical Stage II or III breast cancer
* Clinical Stage II or III NSCLC
* HGSOC, either relapsed after primary treatment, confirmed by biopsy, or suspected on the basis of radiological criteria
* Prostate cancer, with at least one of the following: Gleason Score ≥8, radiologically ≥cT2c, or PSA >10
* Gastric cancer with at least one of the following: Radiological/ecoendoscopic/laparoscopic evidence of node-positive disease, infiltration of the serosa or the surrounding organs, diffuse subtype as histology.

Exclusion Criteria:

* Unable to provide informed consent
* Unable to undergo surgery
* Radiological evidence of metastatic disease
* Unwilling to be subjected to longitudinal plasma samples collection
* Prior diagnosis of a malignant tumor for which the patients underwent any type of anti-neoplastic treatment within 2 years prior to the study screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2033-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
ctDNA detection after surgery | 28 days
  To determine the rate of ctDNA detection after surgery (≤28 days) as a feasibility endpoint;
ctDNA detection at 6 months after the start of adjuvant therapy | 6 month
  To determine the rate of ctDNA detection at 6 months following the initiation of adjuvant therapy in the overall study population.

SECONDARY OUTCOMES:
ctDNA detection at 6 months vs baseline | 6 months
  Evaluate the rate of ctDNA detection at 6 months following the start of adjuvant therapy, stratified by baseline ctDNA status (positive vs negative) and tumor type
ctDNA detection end of adjuvant therapy | up to 8 years
  To evaluate the rate of ctDNA detection at the planned end of adjuvant therapy, as per standard protocol by tumor type
ctDNA detection at 6 months and 12-month, 24-month, and 36-month | 36-month recurrence-free survival
  To assess the association between ctDNA detection at 6 months and 12-month, 24-month, and 36-month recurrence-free survival
ctDNA detection and radiological diagnosis of metastatic disease | up to 8 years
  To analyze the lead time between ctDNA detection and radiological diagnosis of metastatic disease in patients who experience recurrence
Lack of ctDNA clearance | up to 8 years
  To identify genomic and transcriptomic alterations in the primary tumor associated with a lack of ctDNA clearance at landmark analyses
Likelihood of ctDNA clearance and recurrence risk | up to 8 years
  To develop an AI-based prediction model, leveraging multi-omic data and whole slide images of the primary tumor, to predict the likelihood of ctDNA clearance and recurrence risk

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Curigliano, Principal Investigator — European Institute of Oncology; Pier Giuseppe Pelicci, MD, Principal Investigator — European Institute of Oncology; Luca Mazzarella, MD, Principal Investigator — European Institute of Oncology; Antonio Marra, MD, Principal Investigator — European Institute of Oncology

IPD SHARING:
Plan to Share IPD: Undecided